CLINICAL TRIAL: NCT01343862
Title: The Effect of Single Dose D-Cycloserine on Cognitive Outcome in Moderate TBI Patients
Brief Title: The Effect of Single Dose D-Cycloserine on Cognitive Outcome in Moderate Traumatic Brain Injury (TBI) Patients
Acronym: DCS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Guy Rosenthal, MD, Hadassah-Hebrew University Medical Center, Department of Neurosurgery, Hadassah-Hebrew University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0046-10-HMO
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Traumatic Brain Injury
Keywords: moderate traumatic brain injury; brain contusion
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Contusion | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D- Cycloserine (Experimental)
  Interventions: Drug: D-cycloserine
- sugar pill (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: D-cycloserine — single dose of D-cycloserine given 48-72 hours after moderate traumatic brain injury
  Other Names: seromycin
  Arms: D- Cycloserine
Drug: placebo — A sugar pill will be given to those patients randomized to the control group at 48-72 hours after moderate brain injury
  Arms: sugar pill

SUMMARY:
In this study of patients with moderate traumatic brain injury with frontal brain contusions patients will be randomized to treatment with a single dose of either D-cycloserine or placebo given 48-72 hours after injury.

Patients will undergo intensive neurocognitive testing at 3 and 6 months after injury to assess whether treatment with a single dose of D-cycloserine improves cognitive outcome after moderate brain injury.

ELIGIBILITY:
Inclusion Criteria:

1. TBI diagnosed by history and/or clinical examination with presenting GCS between 9 -13
2. Age between 18 and 55 years
3. Frontal cerebral contusion(s) located in the frontal cortex and/or traumatic subarachnoid hemorrhage on initial CT scan
4. Prior to randomization, patient is able to swallow an orally administered tablet or has a nasogastric tube in place per medical indication
5. Informed consent will be obtained in those patients who have regained full cognition and judgment following their injury and are fully capable of understanding the study protocol, its risks and potential benefits, and of giving informed consent for participation in the study. In any patient that has not regained full cognition and judgment, only a temporary legal guardian (apotropos) appointed by an authorized judge that has been given a full explanation of the study protocol, its risks and potential benefits will be authorized to give informed consent for participation in the study.

Exclusion Criteria:

1. Penetrating brain injury
2. Any traumatic intracranial lesion requiring neurosurgical intervention prior to time of randomization
3. Other severe systemic injuries leading to severe hypotension, hemodynamic instability following initial resuscitation (SBP < 90 mmHg), severe hypoxia.
4. Intubation lasting > 12 hours prior to randomization
5. Suspected or confirmed pregnancy or lactating women
6. Any spinal cord injury
7. Known or CT scan evidence of previous major cerebral damage
8. Any severe concomitant condition (malignancy, renal, hepatic, or major psychiatric disorder)
9. Known treatment with another investigational drug within 30 days of injury
10. Known contraindication to enteral administration of drug prior to randomization (GI bleed, ileus, severe abdominal injury, etc.)
11. Known contraindication to placement of a nasogastric tube in patients unable to swallow an orally administered tablet

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
A battery of neuropsychological tests at 3 and 6 months post-injury | 3 and 6 months post-injury
  * Symbol Digit Modalities Test (Smith 1973)
  * Trail Making Test (TMT) (Reitan, Hom et al. 1988)
  * Digit Span (DS) from the WAIS-III
  * Rey Auditory Verbal Learning Test (RAVLT) (Rey 1955; Lezak 2004)
  * Wisconsin Card Sorting Test (WCST) (Psychological Assessment Resources. Computerised Wisconsin Card Sort Task Version 4 (WCST). Psychological Assessment Resources; 2003).
  * Test of Variables of Attention (TOVA) (Test of Variables of Attention: Clinical Manual. Los Alamitos: The TOVA Company).
  * Behavioral Assessment of the Dysexecutive Syndrome (BADS) (Erez, Rothschild et al. 2009)

SECONDARY OUTCOMES:
Glasgow Outcome Score - Extended (GOS-E) | 3 and 6 months post injury

CONTACTS AND LOCATIONS:
Overall Officials: Guy Rosenthal, MD, Principal Investigator — Hadassah Medical Organization
Locations (3):
- Israel (3):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan